CLINICAL TRIAL: NCT01904955
Title: Should Colorectal Cancer Patients be Followed After Five Years? Study of Recurrence in a Population Cohort
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Faivre PHRC K 2010
Record Dates: First submitted 2013-07-08; First posted 2013-07-22 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2013-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

SUMMARY:
The results of this study will make it possible, thanks to better understanding of the natural history of colorectal cancer, to define new treatment and surveillance strategies for colorectal cancers resected with curative intent, so as to improve management and thus improve patient survival.

These data will also make it possible to calculate the prevalence of patients who require treatment or surveillance because of their disease.

ELIGIBILITY:
Inclusion Criteria:

* with adenocarcinoma of the colon or rectum (ICD-O: C18, C19 and C20)
* residing in the département of Côte-d'Or (501,000 inhabitants according to the 1999 census) or Calvados (511, 012 inhabitants) at the moment of diagnosis
* recorded by either Registry between January 1985 and December 2000
* treated by resection with a curative intent.

Exclusion Criteria:

Will be excluded other morphologic tumours and initially metastatic colorectal cancers, anal cancers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with adenocarcinoma of the colon or rectum
Sampling Method: Probability Sample
Enrollment: 598 (Actual)
Dates: Start 2010-09; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
data concerning evolving relapse | during the 10 years following resection for colorectal cancer with curative intent
  * the date of recurrence
  * the site
  * the finality of the surgical treatment (resection with curative intent defined as macroscopically complete resection, without involvement of the surgical margin in the histological examination)
  * the non-surgical adjuvant or palliative treatments (radiotherapy, chemotherapy).

CONTACTS AND LOCATIONS:
Overall Officials: FAIVRE Jean, Principal Investigator — CHU Dijon Gastroentérologie
Locations (1):
- CHU de Dijon, Dijon, France